CLINICAL TRIAL: NCT00007033
Title: Study of Magnesium Sulfate in Children With Reduced Bone Density Secondary to Chronic Cholestatic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other)
Purpose: Treatment
Other Study IDs: 199/15488; CHMC-C-91-3-7
Record Dates: First submitted 2000-12-06; First posted 2000-12-07 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2002-04

CONDITIONS: Alagille Syndrome; Cholestasis; Biliary Atresia
Keywords: Alagille syndrome; biliary atresia; cholestasis; gastrointestinal disorders; rare disease
MeSH Terms: conditions — Alagille Syndrome; Cholestasis; Biliary Atresia; Gastrointestinal Diseases; Rare Diseases | interventions — gluconic acid; Magnesium Sulfate

INTERVENTIONS:
Drug: magnesium gluconate
Drug: magnesium sulfate

SUMMARY:
OBJECTIVES:

I. Determine the role of magnesium deficiency in the pathogenesis of decreased serum vitamin D and reduced bone density in children with chronic cholestatic liver disease.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive magnesium sulfate IV over 1 hour on day 3. Patients then receive oral magnesium gluconate supplementation daily. Treatment with magnesium sulfate repeats once at 3-6 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of liver disease with chronic cholestasis Nonsyndromic intrahepatic cholestasis Alagille's syndrome Extrahepatic biliary atresia
* Direct bilirubin greater than 2 mg/dL OR Bile acids greater than 20 micromoles/L
* No hepatic decompensation defined as one or more of the following: Ascites Peripheral edema PT at least 4 seconds longer than control Albumin less than 3 g/dL

--Patient Characteristics--

* Renal: No significant renal disease
* Cardiovascular: No significant cardiovascular disease
* Pulmonary: No significant pulmonary disease

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25
Dates: Start 2000-10

CONTACTS AND LOCATIONS:
Overall Officials: James Heubi, Study Chair — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Children's Hospital Medical Center - Cincinnati, Cincinnati, Ohio, United States

REFERENCES:
- [Result] Heubi JE, Wiechmann DA, Creutzinger V, Setchell KD, Squires R Jr, Couser R, Rhodes P. Tauroursodeoxycholic acid (TUDCA) in the prevention of total parenteral nutrition-associated liver disease. J Pediatr. 2002 Aug;141(2):237-42. doi: 10.1067/mpd.2002.125802. PMID 12183720